CLINICAL TRIAL: NCT01409057
Title: SEOPCAB: Effect of Heart-lung-machine on Selenium Status of Cardiac Surgical Patients Undergoing Coronary Bypass Surgery
Brief Title: Effect of Heart-lung-machine on Selenium Status of Cardiac Surgical Patients Undergoing Coronary Bypass Surgery
Acronym: SEOPCAB
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A 10-086 SEOPCAB
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Selenium Level
Keywords: Inflammation parameters; Various blood values; Clinical Outcome; Residence in ICU/ Hospital; SAPS-Score; SOFA-Score; Duration of artificial respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No heart lung machine: Coronary-artery-disease
- Heart lung machine: Coronary artery disease

SUMMARY:
Since selenium has demonstrated significant characteristics for a series of biochemical processes, for antioxidant activity and immune stimulation, this observational study should represent the effect of heart-lung-machine on selenium status of cardiac surgical patients undergoing coronary bypass surgery. It will be examined in (approximately 100) adult patients, under which 50 patients are operated conventionally (meaning with the use of heart-lung-machine). Another 50 patients are operated on beating heart without the use of heart-lung-machine (OPCAB = "off pump coronary artery bypass"). The allocation of individual patients in these two groups is done according to clinical criteria and is undertaken by the operating surgeon.

DETAILED DESCRIPTION:
To produce two comparable groups of patients, the characteristics are recorded using EURO-Score; additionally the groups are "matched" (Matched-Pairs-Analysis).

All patients are operated by the same surgeon (senior physician Dr. A.K. Menon) under general anaesthesia through median sternotomy with elective or urgent indications.

After induction of anaesthesia, within the first hour after admission to the Intensive Care Unit (ICU) and every further morning in the ICU or Intermediate Care Station (IMC), 10ml blood are removed by a central venous catheter, allowing to measure blood selenium levels in whole blood by electrothermal atomic absorption spectrometry.

All blood draws will be held on vascular access, which is lying independently of the study participation for surgery or for intensive care treatment. The blood samples will be stored until completion of the study and its evaluation (up to 24 months) and are discarded afterwards. All data collected are recorded on a documentation sheet.

ELIGIBILITY:
Inclusion Criteria:

* Coronary-3-vessel-disease
* Written informed consent
* Age of 18 years or older
* Study inclusion at the latest on the last evening before surgery

Exclusion Criteria:

* Other serious cardiac diagnosis (i.e. aneurysm, valvular-diseases)
* ischemic cardiomyopathy
* Patients not capable of consenting
* Pregnant or lactating women, women of child-bearing potential in whom pregnancy can not be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 adult patients (male and female), capable of consenting, undergoing cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Perioperative serum levels of selenium | 48 hours
  Perioperative serum levels of selenium in patients undergoing either conventional cardiac surgery with the use of cardiopulmonary-bypass (CPB) or without use of CPB on beating heart.
Perioperative serum levels of macrophage migration inhibitory factor (MIF) | 48 hours
  Perioperative serum levels of macrophage migration inhibitory factor (MIF)in patients undergoing either conventional cardiac surgery with the use of cardiopulmonary-bypass (CPB) or without use of CPB on beating heart.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Rex, Dr. med., Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Derived] Stevanovic A, Coburn M, Menon A, Rossaint R, Heyland D, Schalte G, Werker T, Wonisch W, Kiehntopf M, Goetzenich A, Rex S, Stoppe C. The importance of intraoperative selenium blood levels on organ dysfunction in patients undergoing off-pump cardiac surgery: a randomised controlled trial. PLoS One. 2014 Aug 13;9(8):e104222. doi: 10.1371/journal.pone.0104222. eCollection 2014. PMID 25118980